CLINICAL TRIAL: NCT05915923
Title: Effect of Transcranial Magnetic Stimulation on Dynamic Cerebral Autoregulation in Healthy Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yi Yang (Other)
Responsible Party: Sponsor-Investigator, Yi Yang, Vice President of First Hospital of Jilin University, The First Hospital of Jilin University
Organization: The First Hospital of Jilin University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TMSCA-HA
Record Dates: First submitted 2023-05-22; First posted 2023-06-23 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Transcranial Magnetic Stimulation
Keywords: transcranial magnetic stimulation, healthy adults

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low-frequency rTMS Group (Experimental): Healthy adults treated with 1Hz repetitive transcranial magnetic stimulation (rTMS)
  Interventions: Procedure: 1 Hz Repetitive transcranial magnetic stimulation
- High-frequency rTMS Group (Experimental): Healthy adults treated with 10Hz repetitive transcranial magnetic stimulation (rTMS)
  Interventions: Procedure: 10 Hz Repetitive transcranial magnetic stimulation
- Control group (Sham Comparator): The Control group received rTMS with sham transcranial magnetic stimulation (sham-rTMS)
  Interventions: Procedure: Sham Repetitive transcranial magnetic stimulation

INTERVENTIONS:
Procedure: 1 Hz Repetitive transcranial magnetic stimulation — After enrollment, healthy adults received rTMS once a day (stimulation plan: stimulation of M1 region on the dominant hemisphere at 1Hz)
  Arms: Low-frequency rTMS Group
Procedure: 10 Hz Repetitive transcranial magnetic stimulation — After enrollment, healthy adults received rTMS once a day (stimulation plan: stimulation of M1 region on the dominant hemisphere at 10Hz)
  Arms: High-frequency rTMS Group
Procedure: Sham Repetitive transcranial magnetic stimulation — After enrollment, healthy adults received sham-rTMS once a day with the same parameters as the 10 Hz rTMS group, but the coil rotated 90° away from the scalp
  Arms: Control group

SUMMARY:
The purpose of this study is to determine the effect of transcranial magnetic stimulation with different stimulation modes ( 1Hz, 10Hz, sham stimulation ) on cerebral autoregulation.

DETAILED DESCRIPTION:
Current studies have shown that repetitive transcranial magnetic stimulation (TMS) can change the excitability of nerve cells, improve intracerebral artery blood supply, and even reduce the degree of neurological impairment in patients with ischemic stroke.Dynamic cerebral autoregulation (dCA), refers to a complex process in which small intracranial arteries contract or relax to maintain relatively stable cerebral blood volume when systemic arterial blood pressure changes, which can predict the prognosis of patients with ischemic stroke. In this study, we hypothesis that TMS provides neuro-protection by means of improving dCA.

ELIGIBILITY:
Inclusion Criteria:

1. Age≥18 years, < 60 years, both genders；
2. Willing to participate and sign the informed consent；
3. Bilateral temporal windows were well penetrated;

Exclusion Criteria:

1. Complaints of previous or existing chronic organic diseases ( stroke, Parkinson 's disease, hypertension, diabetes, etc. ), mental diseases ( bipolar disorder, personality disorder, schizophrenia, etc. ), or cognitive impairment;
2. Suffering from infectious diseases in late one month;
3. Pregnancy or breast-feeding;
4. Sleep disorders, anxiety and depression,
5. Alcohol or drug abuse;
6. History of prescription drugs or over-the-counter (OTC) drugs in the past 2 weeks;
7. History of epilepsy or family history of epilepsy;
8. Implants ( stents or metals );
9. Other conditions that the researchers think are not suitable for the project.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-08-02 (Actual); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-04-20 (Estimated)

PRIMARY OUTCOMES:
The differences of phase difference (PD) at 30 minutes after transcranial magnetic stimulation under different stimulation modes (1Hz, 10 Hz, sham stimulation). | 0-30minutes
  A cerebral autoregulation parameter derived from transfer function analysis. Continuous cerebral blood flow velocities of bilateral middle cerebral artery will be assessed noninvasively using transcranial Doppler. Spontaneous arterial blood pressure will be simultaneously recorded using a servo-controlled plethysmograph on the left or right middle finger with an appropriate finger cuff size. Transfer function analysis will be used to derive the cerebral autoregulatory parameter.

SECONDARY OUTCOMES:
To compare the difference of phase difference (PD) at 1hour, 6hours and 24hours after transcranial magnetic stimulation under different stimulation modes (1Hz, 10Hz, sham stimulation). | 0-1hour; 0-6hours; 0-24hours
  A cerebral autoregulation parameter derived from transfer function analysis. Continuous cerebral blood flow velocities of bilateral middle cerebral artery will be assessed noninvasively using transcranial Doppler. Spontaneous arterial blood pressure will be simultaneously recorded using a servo-controlled plethysmograph on the left or right middle finger with an appropriate finger cuff size. Transfer function analysis will be used to derive the cerebral autoregulatory parameter.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Hospital of Jilin University, Jilin, China